CLINICAL TRIAL: NCT06495164
Title: Palbociclib Treatment Patterns and Outcomes in HR+/HER2- MBC: Flatiron Database Analysis
Brief Title: A Real-life Study to Understand the Use and Effects of Palbociclib in US Patients With Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481189; NCT06495164 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Malignant Neoplasm of Breast
Keywords: Metastatic breast cancer; CDK4/6 inhibitor; Real-world data; Retrospective observational study; Palbociclib; Overall survival
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Aromatase Inhibitors; Letrozole; Anastrozole; exemestane; ribociclib; abemaciclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Palbociclib + aromatase inhibitor (AI): Oral palbociclib + AI combination treatment regimen as decided by physician
  Interventions: Drug: Palbociclib; Drug: Aromatase inhibitor
- Aromatase inhibitor (AI): Oral AI treatment regimen as decided by physician
  Interventions: Drug: Aromatase inhibitor
- Abemaciclib plus aromatase inhibitor (AI): Oral abemaciclib plus AI treatment regimen as decided by physician
  Interventions: Drug: Palbociclib; Drug: Aromatase inhibitor; Drug: Abemaciclib
- Ribociclib plus aromatase inhibitor (AI): Oral ribociclib plus AI as decided by physician
  Interventions: Drug: Aromatase inhibitor; Drug: Ribociclib

INTERVENTIONS:
Drug: Palbociclib — CDK4/6 inhibitor
  Other Names: Ibrance
  Groups: Abemaciclib plus aromatase inhibitor (AI); Palbociclib + aromatase inhibitor (AI)
Drug: Aromatase inhibitor — Aromatase inhibitor
  Other Names: a class of drugs included in the study: letrozole (Femara), anastrozole (Arimidex), and exemestane (Aromasin)
Drug: Ribociclib — CDK4/6 inhibitor
  Other Names: Kisqali
  Groups: Ribociclib plus aromatase inhibitor (AI)
Drug: Abemaciclib — CDK4/6 inhibitor
  Other Names: Verzenio
  Groups: Abemaciclib plus aromatase inhibitor (AI)

SUMMARY:
Palbociclib, the first oral CDK4/6 inhibitor, is an approved medicine indicated for the treatment of a kind of advanced/metastatic breast cancer (MBC), called hormone receptors positive (HR+)/ Human epidermal growth factor receptor 2 negative (HER2-) disease. Palbociclib is given orally in combination with hormonal therapies.

The purpose of this study is to better understand how Palbociclib combination is used in real-life conditions and its clinical impact compared with hormonal therapy. The study will also evaluate how long patients take the different CDK 4/6 inhibitor drugs and whether using those drugs impacts the use of chemotherapy later.

Male and female patients aged 18 years old or more presenting the following conditions will be selected for the study:

* HR+/HER2- MBC
* First treatment with Palbociclib, hormonal therapy, or other CDK4/6 inhibitors after MBC diagnosis The study will use data without personal identity, which were obtained from medical records in routine clinical practice.

ELIGIBILITY:
Patients are eligible for the study if they were 18 years of age or older at MBC diagnosis, had HR+/HER2- confirmed and initiated first line therapy (CDK4/6i, ET, CT, or other) in the metastatic setting during the period from February 2015 through June 2022 or data cutoff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Flatiron Health Database is a longitudinal, demographically, and geographically diverse dataset derived from EHR data from over 280 cancer clinics (~800 sites of care) including more than 3.0 million active US cancer patients available for analysis. This study uses secondary de-identified Flatiron Health data that involve men and women who had been diagnosed with HR+/HER2-MBC in the United States.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From start of index line of therapy to death, February 2015 - December 2022 or data cutoff

SECONDARY OUTCOMES:
Real Progression Free Survival (rwPFS) | From start of index line of therapy to death or disease progression, February 2015 - December 2022 or data cutoff
Progression Free Survival 2 | from start of index treatment to disease progression on the 2nd line of therapy or death, February 2015 - December 2022 or data cutoff
Real-World Tumor Response (rwTR) | From start of index treatment to tumor response, February 2015 - December 2022 or data cutoff
Duration of treatment | from index treatment initiation to end of the treatment, February 2015 - December 2022 or data cutoff
Time to chemotherapy | from index treatment initiation to subsequent chemotherapy, February 2015 - December 2022 or data cutoff

OTHER OUTCOMES:
Early discontinuation | from index treatment initiation to discontinuation between February 2015 - December 2022 or data cutoff
Dose adjustment | from index treatment initiation to initial dose change, February 2015 - December 2022 or data cutoff

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Lynce F, Liu X, Li B, McRoy L, Chen C, Liu R, Rugo HS. Real-world effectiveness of palbociclib plus an aromatase inhibitor in HR+/HER2- MBC patients living in disadvantaged neighborhoods. NPJ Breast Cancer. 2025 Jul 21;11(1):75. doi: 10.1038/s41523-025-00786-z. PMID 40691446
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481189